CLINICAL TRIAL: NCT02837692
Title: An Open-Label Single Dose Study to Assess the Effects of Age and Gender on the Pharmacokinetics of JNJ-42847922 in Healthy Adults
Brief Title: A Study to Assess the Effects of Age and Gender on the Pharmacokinetics of JNJ-42847922 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108176; 42847922EDI1014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-06-02; First posted 2016-07-19 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants assigned to Cohort 1 group A (elderly non-Asian), group B (young healthy non-Asian) and group C (healthy Japanese) will receive JNJ-42847922 10 mg, 3 hours after completing dinner.
  Interventions: Drug: JNJ-42847922 10 milligram (mg)
- Cohort 2 (Experimental): Participants assigned to Cohort 2 group A, group B and group C will receive JNJ-42847922 20 mg, 3 hours after completing dinner.
  Interventions: Drug: JNJ-42847922 20 mg
- Cohort 3 (Experimental): Participants assigned to Cohort 3 group A and group C will receive JNJ-42847922 40 mg, 3 hours after completing dinner. Participants in group B will receive JNJ-42847922 40 mg, 3 hours after completing dinner in Period 1, followed by at least 7 days washout period, further followed by JNJ-42847922 40 mg, immediately after completing dinner.
  Interventions: Drug: JNJ-42847922 40 mg
- Cohort 4 (Experimental): Participants assigned to Cohort 4 group B will receive JNJ-42847922 60 or 80 mg, 3 hours after completing dinner.
  Interventions: Drug: JNJ-42847922 60 or 80 mg

INTERVENTIONS:
Drug: JNJ-42847922 10 milligram (mg) — JNJ-42847922 will be administered as single tablet of 10 mg, orally, once on Day 1.
  Arms: Cohort 1
Drug: JNJ-42847922 20 mg — JNJ-42847922 will be administered as 1 tablet of 20 mg, orally, once on Day 1.
  Arms: Cohort 2
Drug: JNJ-42847922 40 mg — JNJ-42847922 will be administered as 2 tablets of 20 mg, orally, once on Day 1.
  Arms: Cohort 3
Drug: JNJ-42847922 60 or 80 mg — JNJ-42847922 will be administered as 3 or 4 tablets of 20 mg, orally, once on Day 1. Dose to be determined from Cohort 3, Period 1.
  Arms: Cohort 4

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of single-dose evening administration of JNJ-42847922 in elderly non-Asian adults compared with weight- and gender-matched young healthy non-Asian adults and to assess the pharmacokinetics of single-dose evening administration of JNJ-42847922 in healthy Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

* In Group A: For each cohort, 10 elderly non-Asian adults greater than or equal to (>=)65 years old, with at least 2 participants >=70 years and <75 years old, at least 2 participants >=75 years old, with 5 participants of each sex; In Group B: For each cohort, 10 young healthy non-Asian adults 18 to 45 years old, inclusive, matched to elderly participants in the same cohort by gender and body weight (plus [+] or minus [-]5 kilogram [kg]); In Group C: For each cohort, 10 healthy Japanese adults 20 to 60 years old, inclusive, who have resided outside of Japan for less than or equal to (<=)10 years, have parents and maternal and paternal grandparents who are Japanese, who primarily consume a Japanese diet, with 5 participants of each sex
* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Group B and Group C: If a woman, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day 1 of the treatment period
* Group B and Group C: If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 3 months after the last study drug administration
* If a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Has body mass index (BMI) (weight kilogram[kg]/height^2 meter[m]^2) between 18 and 30 kg/m2 (inclusive) with a body weight not less than 50 kg for non-Asian subjects (Group A and Group B) and not less than 45 kg for Japanese subjects (Group C)

Exclusion Criteria:

* Received a known inhibitor of cytochrome P450 3A4 (CYP3A4) or CYP2C9 activity within 28 days or a period less than 5 times the drugs half-life; whichever is longer, before the first dose of the study drug is scheduled
* Consumption of products containing grapefruit or Seville oranges within 28 days before the first dose of the study drug is scheduled
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-42847922 | Day 1 (Pre-dose) up to Day 3
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) of JNJ-42847922 | Day 1 (Pre-dose) up to Day 3
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-42847922 | Day 1 (Pre-dose) up to Day 3
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events as a measure of safety and tolerability | Baseline up to 10 days after last dose of study drug (Day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Cypress, California
  - Knoxville, Tennessee